CLINICAL TRIAL: NCT01610817
Title: Impact of a Procedure for the Information and Active Participation of the Patient in the Primary Care Prescription of Antihypertensives : InPAct Study (Information for Participating Actively in Cardiovascular Treatment)
Brief Title: Impact of a Procedure for the Information and Active Participation of the Patient in the Primary Care Prescription of Antihypertensives
Acronym: InPAct
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50802; PHRC National 2011 (Other: government)
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Patients on Anti-hypertensive Medication
Keywords: Patient information and active participation; Patient safety; Health education; Adverse drug event; Primary care; Antihypertensive drugs
MeSH Terms: conditions — Health Education; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with the InPAct intervention: The InPAct intervention will be presented to the last patients recruited by each general practitioner
  Interventions: Other: InPAct : Information for Participating Actively in cardiovascular treatment
- Patients without the InPAct intervention: The InPAct intervention will not be presented to the first patients recruited by each general practitioner

INTERVENTIONS:
Other: InPAct : Information for Participating Actively in cardiovascular treatment — Educational guide presented by general practitioners to the patients. A first part of the guide contains some information on cardiovascular risk and on the benefits and risks of antihypertensive drugs. A second part of the guide consists of encouraging the patient to take an active part in monitoring of its treatment.
  Groups: Patients with the InPAct intervention

SUMMARY:
Adverse drug events (ADEs) are responsible for 3.6% of the hospitalisations in France. 50% of these ADEs could be preventable. Cardiovascular drugs are frequently involved in ADEs. A common underlying factor of such events is inadequate communication between patients and medical personnel. General practitioners (GP) often initiate the treatment of hypertension, being generally the first prescribers of these medications. 12.6% of the patients present an ADE with hypertensive drug after 3 months. The InPAct procedure is a tool to facilitate communication in order to improve patient safety in primary care. In the context of the primary care prescription of an antihypertensive drug, the GP informs the patient about hypertension, cardiovascular risk, and the benefits and risks of antihypertensive drugs, which helps the patient to detect and declare situations involving a heightened risk of antihypertensive-related ADEs. The aim of the InPAct study is to evaluate the efficiency of the InPAct intervention in primary care.

DETAILED DESCRIPTION:
A stepped wedge cluster randomized study, with 8 clusters and 5 periods of 3 months each. Each cluster is composed of about ten general practitioners. The InPAct intervention will not be presented to the first patients recruited by each general practitioner, whereas it will be presented to all their last patients. The period of intervention introduction by each general practitioner will be randomized amongst the 5 periods.

ELIGIBILITY:
Inclusion Criteria:

* Patient monitored for essential hypertension requiring a first prescription, a renewal or a change of antihypertensive drug treatment
* Patient with the ability to understand and express themselves in French
* Patient accepting to communicate his phone number and accepting a telephone survey within the fourth month following its inclusion in the study.

Exclusion Criteria :

* Patient with a psychiatric disorder or a progressive dementia.
* Patient with hypertension in pregnancy or secondary hypertension.
* Patient with an acute hypertensive crisis.
* Patient under guardianship.
* Patient who is likely to move or may have an irregular follow up within 6 months following its inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients on anti-hypertensive medication. Patients of 85 general practitioners selected in Rhone-Alps/Auvergne and Paris region in France.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients on antihypertensive drug reporting themselves at least one Adverse Drug Event (ADE) to their general practitioner during their 90 days of follow up. | During the study : 19 months
  Symptoms could have begun before patient inclusion in the study, but symptoms have to be related to an ADE and reported during the 90 days of patient follow up.

SECONDARY OUTCOMES:
The proportion of patients on antihypertensive drug with at least an ADE detected (reported by the patient himself, or not) during their 90 days of follow up. | During the study : 19 months
  Symptoms could have begun before patient inclusion in the study, but symptoms have to be related to an ADE during the 90 days of patient follow up.
The proportion of patients on antihypertensive drug presenting at least one situation of risk for ADE during the 90 days of patient follow up. | During the study : 19 months
The proportion of patients on antihypertensive drug for whom a physician has changed or modified at least one prescription during the 90 days of patient follow up. | During the study : 19 months
  This modification had to be made following an ADE or a situation of risk for ADE associated with taking an anti-hypertensive drug or a drug associated with antihypertensive treatment.
The proportion of patients who developed at least one complication following an ADE detected during the 90 days of patient follow up. | During the study : 19 months
A mean score of patient satisfaction regarding the communication and information on drug prescription and management of hypertension by the general practitioner, during the 90 days of patient follow up. | During the study : 19 months
A mean score of patient skill in health after 90 days of follow-up, including a score of patient knowledge on cardiovascular risk and on the benefits and risks of antihypertensive drugs, and a score of patient skill in situation of ADE. | During the study : 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille COLIN, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Buchet-Poyau K, Occelli P, Touzet S, Langlois-Jacques C, Figon S, Dubois JP, Duclos A, Chaneliere M, Colin C, Rabilloud M, Keriel-Gascou M. Improving patient self-reporting of antihypertensive adverse drug events in primary care: a stepped wedge cluster randomised trial. BMC Fam Pract. 2021 Aug 7;22(1):165. doi: 10.1186/s12875-021-01478-w. PMID 34364386
- [Derived] Keriel-Gascou M, Buchet-Poyau K, Duclos A, Rabilloud M, Figon S, Dubois JP, Brami J, Vial T, Colin C. Evaluation of an interactive program for preventing adverse drug events in primary care: study protocol of the InPAct cluster randomised stepped wedge trial. Implement Sci. 2013 Jun 19;8:69. doi: 10.1186/1748-5908-8-69. PMID 23782470